CLINICAL TRIAL: NCT02245594
Title: Gastrointestinal Motility and Sleep Disturbances in Patients With Quiescent Crohn's Disease
Brief Title: GI Symptoms and Sleep Disturbances in Patients With Quiescent Crohns Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: MbCrohnRemission+Symp
Record Dates: First submitted 2014-09-08; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease; Sleep Disturbances
Keywords: Gastrointestinal motility; Motility Tracking System (MTS); Transit time; Sleep pattern
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A single blood sample (TNF-α, IL-1, IL-6) will be taken at the laboratory.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gl motility and sleep pattern

SUMMARY:
In this study we would like to clarify the effect of long lasting Crohn's Disease on motility of the gastrointestinal system in patient and the effect regarding sleep disturbances. This will be done with a newly developed 3D-Motility-and-Transit-detector (Motilis Medica, Schweiz) and the well known polysomnographic equipment.

Our hypothesises are:

Patients with ileocoecal and/or colonic CD in remission and gastrointestinal symptoms have abnormal colonic transit (primary endpoint).

1. Patients with ileocoecal and/or colonic CD in remission and gastrointestinal symptoms have abnormal gastric emptying and small intestinal transit (secondary endpoints).
2. Total and segmental transit times found in patients with CD will be compared with corresponding transit times in healthy volunteers found in a previous study.
3. Patients with ileocoecal and/or colonic CD in remission have abnormal sleep patterns.
4. Nocturnal basic colonic activity, have changed in patients with ileocoecal and/or colonic CD in remission and sleep disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD based on accepted endoscopic and histological criteria (according to ECCO guidelines (17) )
* Age ≥18 years
* A minimum disease duration of five years
* Remission defined by Faecal calprotectin < 100 and CRP level within normal values for a minimum of 1 month
* Baseline values:

  * CRP normal
  * Faecal calprotectin < 100
* Ileocoecal and/or colic localization of disease (Montreal phenotype classification)
* One or more IBS-like-symptoms (abdominal pain and discomfort, diarrhea, constipation)

Exclusion Criteria:

* Stricturizing CD
* Obvious stenotic symptoms
* Previous major gastrointestinal surgery
* Diagnosis of other gastrointestinal diseases affecting motility (ex. Coeliac disease)
* Medication altering gastrointestinal motility
* Hepatobiliary disease (PSC)
* Diabetes Mellitus
* Metabolic disorder
* Bacterial overgrowth (hydrogen breath test)
* Planned MR scan in the four weeks following capsule intake (safety precaution)
* Abdominal diameter > 140 cm
* Implanted electronic devices (pacemaker, ICD, etc.)
* Diagnosed sleep disorder
* Pregnancy and breast feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with quiescent Crohn's disease who still have gastrointestinal complaints.Found in the out-patient clinic at Department V (Gastroenterology and Hepatology).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Total and segmental gastrointestinal transit time in patients suffering from CD | Expected average total transit time less than two days, analyzed after 2-3 days
Abnormal sleep pattern in patients with ileocoecal and/or colonic CD in remission | Recorded during a single night, analyzed one of the two following days.

SECONDARY OUTCOMES:
Gastric emptying in CD patients | Less than 1 day, analyzed after 1-3 days
Small intestinal transit time in CD patients | Less than 2 days, analyzed after 2-3 days
Segmental colonic transit time in CD patients | Average less than 2 day, analyzed after 2-3 days
Nocturnal basic colonic activity in patients with ileocoecal and/or colonic CD in remission and sleep disturbances | Recorded during one night, analyzed one of the two following days

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Krogh, MD, Dr. Med, Study Director — Department of Gastroenterology and Hepatology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Gastroenterology and Hepatology, Aarhus C, Denmark